CLINICAL TRIAL: NCT03937193
Title: Normal Range of Superior Mesenteric Artery on Computerized Tomography in Young Chinese Population and Its Correlation With Retroperitoneal Adipose Tissue
Brief Title: Normal Range of Superior Mesenteric Artery in Young Chinese Population and Its Correlation With Retroperitoneal Adipose Tissue
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: North District Hospital (Other)
Responsible Party: Principal Investigator, Professor Winnie W.C. Chu, Professor, Chinese University of Hong Kong
Other Study IDs: 2019.310
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Aortomesenteric Angle; Aortomesenteric Distance; Retroperitoneal Adipose Tissue
Keywords: aortomesenteric angle; aortomesenteric distance; retroperitoneal adipose tissue; computerized tomography; young Chinese population
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-SMAS group: subjects in this group are not clinically diagnosed as superior mesenteric artery syndrome(SMAS).
  Interventions: Diagnostic Test: computerized tomography
- SMAS group: subjects in this group are clinically diagnosed as superior mesenteric artery syndrome(SMAS).
  Interventions: Diagnostic Test: computerized tomography

INTERVENTIONS:
Diagnostic Test: computerized tomography — abdomen contrast computerized tomography performed for both emergency and elective purposes in HK public hospitals.

SUMMARY:
In literature, superior mesenteric artery (SMA) angle, also named as aortomesenteric angle (AMA), varies greatly in both adult and children; while the aortomesenteric distance also ranges widely. Both AMA and AMD are influenced by retroperitoneal fat. Decrease of AMA and AMD may lead to the superior mesenteric artery syndrome(SMAS), which is a rare medical condition mainly presenting with duodenum obstruction. To our knowledge, normal range of AMA and AMD in local young Chinese population remain unclear; on the other hand, there have only a few studies exploring the relationship between them. This project proposes to establish the normal range of AMA and AMD in local young Chinese population, and to further investigate how the retroperitoneal adipose tissue correlates with AMA and AMD. The normal range obtained in this proposed study will provide more specific reference value to distinguish abnormal AMA and AMD, and to improve the diagnosis accuracy of SMAS in local population. Moreover, this study will provide deeper insight concerning the impact of retroperitoneal fat on AMA and AMD.

ELIGIBILITY:
Inclusion Criteria:

* With age range of 10-35 years old.
* Chinese ethnicity.
* With abdomen contrast CT.

Exclusion Criteria:

* Any patients with diagnosis of SMAS will be excluded from the Non-SMAS group.
* Patients who had undergone more than one CT scan during the research period.
* Previous retroperitoneal, abdominal surgery.
* Conditions causing significant weight loss, e.g. anorexia nervosa, malabsorption.
* Presence of abdominal masses or pathology that will affect the anatomy of aorta- superior mesenteric artery and the retroperitoneal structures.
* Presence of severe scoliosis and/or history of spinal fixation that may increase incidence of SMA syndrome.
* Presence of free intraperitoneal or retroperitoneal fluid that may affect fat measurement, e.g. following trauma, or ascites.

Ages: 10 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: The investigators will retrospectively recruit individuals from the local population who had undergone abdomen contrast CT scans within hospitals in the New Territories East Cluster (NTEC) of Hong Kong for both emergency and elective purposes in the year 2013-2019. Total sample will comprise two groups: (1) Non-SMAS Group (N=500); and (2) SMAS group (N=10).
Sampling Method: Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
aortomesenteric angle (AMA) | 2 years
  aortomesenteric angle in degree measured on sagittal CT image
aortomesenteric distance (AMD) | 2 years
  aortomesenteric distance in millimeter(mm) on axial CT image
visceral fat area | 2 years
  visceral fat area in square centimeter(cm2) evaluated by image post-processing software
subcutaneous fat area | 2 years
  subcutaneous fat area in square centimeter(cm2) evaluated by image post-processing software
area ratio of visceral fat to subcutaneous fat | 2 years
  area ratio in percentage(%)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ho Yam, MBChB, Principal Investigator — Department of Radiology, North District Hospital, Hong Kong
Locations (1):
- Department of Radiology， North District Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No